CLINICAL TRIAL: NCT03628443
Title: Cardiorenal Risk Stratification Pilot Study (CRiSPS): Using FGF-23 as a Risk Stratification Biomarker in Patients With Heart Failure and Chronic Kidney Disease as a Predictor of 1-year Morbidity and Mortality Risk
Brief Title: Cardiorenal Risk Stratification Pilot Study
Acronym: CRiSPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coney Island Hospital, Brooklyn, NY (Other)
Responsible Party: Principal Investigator, George Juang, Cardiology Fellowship Program Director, Coney Island Hospital, Brooklyn, NY
Other Study IDs: 18-08-172-378(HHC)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cardio-Renal Syndrome; Heart Failure; Chronic Kidney Diseases
Keywords: CKD; HFrEF; HFpEF; FGF23; Dialysis; Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Cardio-Renal Syndrome; Heart Failure; Renal Insufficiency, Chronic; Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood in EDTA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure without Chronic Kidney Disease: This group has patients managed with all types of heart failure without concomitant chronic kidney disease.
  Interventions: Diagnostic Test: Fibroblast Growth Factor 23
- Heart Failure with Chronic Kidney Disease: This group has patients managed with all types of heart failure with concomitant chronic kidney disease, without evidence of sustained hyperphosphatemia.
  Interventions: Diagnostic Test: Fibroblast Growth Factor 23

INTERVENTIONS:
Diagnostic Test: Fibroblast Growth Factor 23 — A sample of blood is tested for levels of fibroblast growth factor 23

SUMMARY:
This is prospective cohort study with the purpose of improving our understanding of morbidity and mortality risk in patients with heart failure and chronic kidney disease.

DETAILED DESCRIPTION:
The CDC reports that approximately 5.7 million adults in the U.S. have heart failure (HF), and NHANES reports that 26% of individuals 60 years-of-age and older have Chronic Kidney Disease. NHANES also reports that End-Stage Kidney Disease (ESKD) accounts for $40 billion in Medicare and Non-Medicare costs in 2009; 37% of those patients had a prior episode of HF. These figures demonstrate that the treatment of patients with HF and ESKD costs Americans almost $15 billion annually. A meta-analysis of 16 studies estimates that 63% of HF patients have some kidney impairment; a serum creatinine (Cr)>1.0mg/dL or Glomerular Filtration Rate (GFR)<90 ml/min. Among HF patients with even mildly decreased GFR, mortality increases significantly; those with none, any, and at least moderate CKD experienced a 24%, 38% and 51% 1-year mortality, respectively. In 2015, 66,713 patients were seen at our hospital. About 3% of those patients had a new diagnosis of CHF and at least 30% of those patients diagnosed with CHF had a dual diagnosis of CKD. This population alone accounted for 79,835 of visits in the same year. It is evident that there are both fiscal and ethical incentives, both locally and nationally, to understand how to mitigate disease progression in this population.

Current classification schemes for patients with HF and chronic kidney disease (CKD), cardiorenal syndrome, do not significantly alter management other than managing HF or CKD independently with respect to their individual severity. In CKD, worsening renal function often leads to poor phosphate (PO4) regulation where hyperphosphatemia is significantly associated as a predictor of mortality. Further characterizations of the factors that contribute to hyperphosphatemia implicates Fibroblast Growth Factor 23 (FGF-23) as a major hormone regulator of PO4 levels in the body. FGF-23 has repeatedly demonstrated its use as an independent predictor of mortality in ESKD as well as an independent predictor of worsening renal function in non-diabetic patients with mild CKD. FGF-23 achieves PO4 level control by downregulating PO4 reabsorption via transporters in kidney's proximal tubules as well as the small intestines through an incompletely understood mechanism. This action allows the increased filtration of PO4 without proximal tubule reabsorption as well as indirectly decreased uptake of dietary PO4. In ESKD, the PO4-lowering effects of FGF-23 diminish despite rising FGF-23 levels; this indicates that pathologic hyperphosphatemia represents a decompensated state of PO4 regulation. There are studies that suggest FGF-23 is not only implicated in the worsening of CKD, but the pleiotropic effects of FGF-23 remain to be understood as a factor in cardiovascular disease. Increased FGF-23 levels have been associated with left ventricular dysfunction and atrial fibrillation as well as worsening CKD. In one study, not a single patient with Group 5 CKD had an FGF-23 level lower than 40.2ρg/dL, and more than 70% of those patients had and FGF-23 level greater than 66.1ρg/dL.14 Despite this information, it is not currently known how FGF-23 may be used as a predictor of mortality or progression of CKD in patients with cardiorenal syndrome prior to end-stage renal disease. Significant results from this study may provide a predictable classification scheme based on FGF-23 levels that may be employed in future studies to guide treatment evaluation. The prospect of treatment to reduce morbidity and mortality is supported by studies demonstrating that PO4 binders lower FGF-23 levels, even in healthy volunteers. The study proposed here is an early step in evaluating options to reduce the number of patients that progress to ESRD with a parallel step towards a reduction in significant healthcare costs. Participants in this study will only be observed after they have granted their informed consent. There are no significant potential risks posed by this study as blood collected would be from routine lab vials for the participant population. If the study has significant findings, there are immediate benefits to the population studied and the greater society.

Participants after this study will be equipped with more knowledge to help them understand their risk factors and help them make better decisions about their own healthcare. The investigators hope to achieve a better understanding of what levels of FGF-23 are significantly associated with morbidity and mortality in patients with CHF and CKD. This information can help us answer how current clinicians may better stratify the risks of CHF and CKD; translating theoretical disease predictions into a preventative medicine model. The answer to this question may lay the foundation for treatment and prevention option studies based on FGF-23 levels in patients that are not currently on hemodialysis.

We hypothesize (1) that in participants with congestive heart failure and chronic kidney disease who are not on hemodialysis, worsening heart disease or worsening kidney disease is associated with a significantly elevated FGF-23 serum level AND (2) participants with congestive heart failure and chronic kidney disease who are not on hemodialysis, decreased survival is associated with a significantly elevated FGF-23 serum level.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of congestive heart failure

Exclusion Criteria:

* Patients cannot be on hemodialysis at the study onset.
* Patients cannot have hyperphosphatemia defined as persistent serum phosphorus level>4.5mg/dL at study onset.
* Patients cannot be part of another study for the investigational treatment of heart failure or chronic kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Control Arm: People seen in the outpatient setting with congestive heart failure without renal impairment. Study Arm: People seen in the outpatient setting with congestive heart failure that have some form of renal impairment that did not start the study while on hemodialysis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year from sample date
  The occurrence of death
Worsening Renal Function | 1 year from sample date
  Significant, persistently decreased in estimated glomerular filtration rate
Worsening Cardiac Function | 1 year from sample date
  Decreased ejection fraction, newly documented structural abnormality
End-Stage Renal Disease Progression | 1 year from sample date
  Progression of patient's health condition requiring the initiation of hemodialysis

SECONDARY OUTCOMES:
Hospitalizations | 1 year from sample date
  Number of times the patient was hospitalized
Increased Medication Use | 1 year from sample date
  Number of medication changes during observation period, including for comirbidities
Worsening Control of Co-Morbidities | 1 year from sample date
  Progression of other co-morbid conditions including, diabetes, dyslipidemia, and hypertension.
Urgent visits | 1 year from sample date
  Number of times the patient visited the emergency department, urgent care, or walked into clinic.
Myocardial Infarction | 1 year from sample date
  Myocardial infarction diagnosed during the trial period
Coronary Artery Disease | 1 year from sample date
  Coronary artery disease diagnosed during the trial period
Stroke | 1 year from sample date
  Stroke diagnosed during the trial period
Arrhythmia | 1 year from sample date
  Arrhythmia diagnosed during the trial period

CONTACTS AND LOCATIONS:
Overall Officials: George Juang, MD, Principal Investigator — Coney Island Hospital
Locations (1):
- Coney Island Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Executive Summary: Heart Disease and Stroke Statistics--2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):447-54. doi: 10.1161/CIR.0000000000000366. No abstract available. PMID 26811276
- [Background] Smith GL, Lichtman JH, Bracken MB, Shlipak MG, Phillips CO, DiCapua P, Krumholz HM. Renal impairment and outcomes in heart failure: systematic review and meta-analysis. J Am Coll Cardiol. 2006 May 16;47(10):1987-96. doi: 10.1016/j.jacc.2005.11.084. Epub 2006 Apr 24. PMID 16697315
- [Background] Prie D, Friedlander G. Genetic disorders of renal phosphate transport. N Engl J Med. 2010 Jun 24;362(25):2399-409. doi: 10.1056/NEJMra0904186. No abstract available. PMID 20573928
- [Background] Prie D, Urena Torres P, Friedlander G. Latest findings in phosphate homeostasis. Kidney Int. 2009 May;75(9):882-9. doi: 10.1038/ki.2008.643. Epub 2009 Feb 4. PMID 19190675
- [Background] Ferrari SL, Bonjour JP, Rizzoli R. Fibroblast growth factor-23 relationship to dietary phosphate and renal phosphate handling in healthy young men. J Clin Endocrinol Metab. 2005 Mar;90(3):1519-24. doi: 10.1210/jc.2004-1039. Epub 2004 Dec 21. PMID 15613425
- [Background] Bogadel'nikov IV. [State of the kallikrein-kinin system in bacterial poisoning]. Zh Mikrobiol Epidemiol Immunobiol. 1978 Nov;(11):20-5. No abstract available. Russian. PMID 364890
- [Background] Gutierrez OM, Mannstadt M, Isakova T, Rauh-Hain JA, Tamez H, Shah A, Smith K, Lee H, Thadhani R, Juppner H, Wolf M. Fibroblast growth factor 23 and mortality among patients undergoing hemodialysis. N Engl J Med. 2008 Aug 7;359(6):584-92. doi: 10.1056/NEJMoa0706130. PMID 18687639
- [Background] Fliser D, Kollerits B, Neyer U, Ankerst DP, Lhotta K, Lingenhel A, Ritz E, Kronenberg F; MMKD Study Group; Kuen E, Konig P, Kraatz G, Mann JF, Muller GA, Kohler H, Riegler P. Fibroblast growth factor 23 (FGF23) predicts progression of chronic kidney disease: the Mild to Moderate Kidney Disease (MMKD) Study. J Am Soc Nephrol. 2007 Sep;18(9):2600-8. doi: 10.1681/ASN.2006080936. Epub 2007 Jul 26. PMID 17656479
- [Background] Ikee R, Tsunoda M, Sasaki N, Sato N, Hashimoto N. Emerging effects of sevelamer in chronic kidney disease. Kidney Blood Press Res. 2013;37(1):24-32. doi: 10.1159/000343397. Epub 2013 Mar 6. PMID 23486088
- [Background] Liu S, Quarles LD. How fibroblast growth factor 23 works. J Am Soc Nephrol. 2007 Jun;18(6):1637-47. doi: 10.1681/ASN.2007010068. Epub 2007 May 9. PMID 17494882
- [Background] Larsson T, Nisbeth U, Ljunggren O, Juppner H, Jonsson KB. Circulating concentration of FGF-23 increases as renal function declines in patients with chronic kidney disease, but does not change in response to variation in phosphate intake in healthy volunteers. Kidney Int. 2003 Dec;64(6):2272-9. doi: 10.1046/j.1523-1755.2003.00328.x. PMID 14633152
- [Background] Seiler S, Cremers B, Rebling NM, Hornof F, Jeken J, Kersting S, Steimle C, Ege P, Fehrenz M, Rogacev KS, Scheller B, Bohm M, Fliser D, Heine GH. The phosphatonin fibroblast growth factor 23 links calcium-phosphate metabolism with left-ventricular dysfunction and atrial fibrillation. Eur Heart J. 2011 Nov;32(21):2688-96. doi: 10.1093/eurheartj/ehr215. Epub 2011 Jul 6. PMID 21733911
- [Background] Tanaka S, Fujita S, Kizawa S, Morita H, Ishizaka N. Association between FGF23, alpha-Klotho, and Cardiac Abnormalities among Patients with Various Chronic Kidney Disease Stages. PLoS One. 2016 Jul 11;11(7):e0156860. doi: 10.1371/journal.pone.0156860. eCollection 2016. PMID 27400031
- See also: Kidney Disease Statistics for the United States — https://www.niddk.nih.gov/health-information/health-statistics/kidney-disease